CLINICAL TRIAL: NCT06782165
Title: Long-term Follow up of TMJ Surgery and Evaluation of the 6-month Control as a Prognostic Marker.
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Mattias Ulmner, Lecturer, Karolinska Institutet
Other Study IDs: 2024-06070-01
Record Dates: First submitted 2025-01-02; First posted 2025-01-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Temporomandibular Disorders (TMD); Temporomandibular Joint Disc Displacement, With Reduction; Temporomandibular Joint Disc Displacement, Without Reduction
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Arthroscopy; Diskectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgically treated patients due to temporomandibular joint disc displacment: The cohort has already been operated (arthroscopy or discectomy) due to temporomandibular joint disc displacement during the years 2014-2017, then participating in a prospective cohort study mainly focusing on surgical outcome predictors (ethical approval: 2014/622-31/1 and 2014/764-31/2). These patients will now be offered a clinical and radiological examination approximately 10 years postoperative.
  Interventions: Procedure: Arthroscopy & saline irrigation alone; Procedure: Discectomy

INTERVENTIONS:
Procedure: Arthroscopy & saline irrigation alone — Arthroscopic lysis and lavage refers to an arthroscopic procedure where the temporomandibular joint is rinsed with saline solution and where the joint capsule is distended and where adhesions are lysated bluntly
Procedure: Discectomy — Discectomy refers to open temporomandibular joint surgery where the joint disc is completely removed without being replaced.

SUMMARY:
The goal of this clinical trial is to evaluate the long-term outcome of surgical intervention (arthroscopy or discectomy) due to the diagnoses temporomandibular joint disc displacement with or without displacement. The main questions it aims to answer are:

* Does the surgical outcome recorded at the earlier 6-month follow up persist at the long-term follow up approximately 10 years postoperatively?
* How does the radiologically determined degree of joint degeneration change with time in patients that have had joint surgery? Researchers will compare the six-month surgical outcome to the ten-year outcome to see if temporomandibular joint surgery results are stable over time.

Participants with an earlier performed joint surgery will:

* Have a clinical examination approximately ten years postoperatively.
* Have a temporomandibular joint x-ray scan performed (cone-beam computed tomography).

DETAILED DESCRIPTION:
1. BACKGROUND Disc displacement (DD) of the temporomandibular joint (TMJ) is a common condition, reported to affect up to 20-30% of the population. Fortunately, only a minority of the affected experience pain and restricted mandibular movements, which are common reported signs of DD when symptomatic. Primary treatment for TMJ DD is non-surgical interventions such as orthotic splint, physiotherapy, pharmacological therapy, etc., all showing good outcome. If non-surgical management fails, surgical interventions might be considered. There are several reports on arthrocentesis, arthroscopy, and open joint surgery showing good results when treating TMJ DD. Most surgical reports have a follow-up period between 3-24 months and therefore little is known about the long-term outcome. Studies on arthroscopic treatment of the TMJ with the longest follow-up was found to be between 4.4 to 5 years. All these studies were retrospective. One study reporting on the outcome after arthroscopy was performed with a survey sent to 37 patients 10 year postoperative. The situation is almost the same regarding discectomy, with few clinical reports on long-term follow-up (10 years) of the surgical outcome. A 30-year follow-up survey was made on a Swedish patient material in the 1980´s, showing a good outcome.

   Since there is a shortage of clinical studies exploring long-term outcome of arthroscopic and open joint surgery, the aim of this study is to do a clinical investigation of a patient cohort earlier prospectively followed for a period of six months postoperative. The plan is to do follow-ups at approximately 10 and 15 years postoperatively.
2. HYPOTHESIS/RESEARCH QUESTIONS Our hypothesis is that the six-month postoperative outcome is a predictive marker for long-term outcome regarding surgical intervention due to TMJ DD. The outcome will be longitudinally evaluated by maximum mouth opening capacity, patient reported TMJ pain and TMJ disability. This was the original outcome parameters used for this patient cohort earlier investigated. The ethical permit for the earlier studies is (EPN 2014/764-31/2 and 2014/622-31/1) and the patients had their surgery between 2014 and 2017.

   The primary research question is whether the long-term outcome of surgery in patients with TMJ DD (DDwR and DDwoR) might be correlated to the six-month outcome.

   A secondary question is to investigate the long-term outcome of TMJ surgery due to DD.

   Tertiary questions:
   * Do any of the registered pre-operative variables serve as prognostic markers when correlated to the long-term outcome?
   * is the clinical long- or short-term outcome correlated to the radiological outcome?
   * Is the preoperative radiological examination predictive for the surgical outcome in long- or short-term?
   * Can naturally occurring deterioration of the TMJ surfaces be distinguished from earlier or present symptoms?
3. METHODS 3.1. Study design A prospective longitudinal cohort study.

   3.2. Data source/study population

   Please, see eligability below.

   3.3. Exposure/Intervention The exposure was arthroscopy or discectomy performed between the years 2014 and 2017. A follow up visit/control will be performed to assess the subjective and objective outcome of the exposure.

   3.4. Outcome

   Please, see "outcome measures" below,

   3.5. Sample size

   The trial aims at including all patients that had TMJ surgery (arthroscopy or discectomy) participating in two different studies between the years 2014-2017. Power analysis in section 4.

   3.6. Inclusion criteria

   Please, see "eligibility" below.

   3.7. Exclusion criteria

   Please, see "eligibility" below.

   3.8. Data collection

   All eligible patients will receive a letter with information about the project alongside an appointment for investigation of their TMJ status. At the appointment different variables will be collected according to a case record form, see attachment.

   The assessor/-s will be calibrated in accordance with the DC/TMD criteria. The surgeon originally responsible for the surgical treatment of the patients will not be involved in the assessment of the patients, minimizing any potential interviewer's bias.

   Anamnestic data: age, sex, operated joint (left, right), present health issues, present medication, later operation of TMJ (Y/N), use of orthotic splint (Y/N), TMJ exercise (Y/N), painkillers due to TMJ disorder (Y/N), continuous controls at specialist in gnathology (Y/N), continuous controls at physiotherapist (Y/N), patient-reported TMJ disability (VAS 0-10), patient-reported TMJ pain (VAS 0-10), patient-reported psycho-social impairment because of TMJ disorder (VAS 0-10), patient-reported global pain (VAS 0-10).

   Objective data: MIO (mm), lateral excursive movement right and left(mm), protrusion (mm), pain upon palpating masticatory muscles (Y/N), pain upon lateral joint palpation (Y/N).

   3.9. Radiological evaluation

   At the timepoint of examination, a radiological evaluation of the TMJ status will be made with a cone beam computed tomography (CBCT). The patients were evaluated preoperatively with a CBCT scan, which makes it possible to evaluate eventual time dependent deterioration of the joints. The CBCT will be taken according to a strict protocol (the departments usual CBCT examination protocol regarding TMJ will be used): FOV 15cm x 6cm, 90kV, 125mAs, voxel size 0,3cm3. Based on the dose area product (DAP) the resulting/effective radiation dose is 0.2 mSv/examination.

   The preoperative CBCTs and the CBCTs taken at the planned follow-ups will be qualitatively and quantitatively examined regarding hard- and soft-tissue changes in the TMJ area. If there is a sufficient postoperative radiological examination already exposed during the last year, this will be used instead of taking a new CBCT.
4. STATISTICAL ANALYSIS With a power of 90% (β) and α equal to 0.05, 44 patients need to be enrolled to detect a VAS difference of 1 unit (standard deviation: 2). The DDwoR cohort who had arthroscopy consists of 67 patients and should be sufficient for the purpose.

   Preoperative data and surgical outcome will be analysed with ordinal regression to evaluate possible outcome predictors. Repeated measurements as MIO, TMJ pain and TMJ disability will be analysed with mixed effects model. If linear relations between pre- and post-operative values exists, multiplicative linear regression might be used.

   All statistical analyses will be made with STATA/SE 16.1, Statacorp, Texas.
5. TIME PLAN

   The study includes one post-operative control for patients (n=91) who earlier had their TMJs operated. The control will take approximately 30 minutes. The control will be scheduled in 2025. The gathered information will be analysed 2026 and a manuscript produced and submitted during 2027.
6. ETHICS

   The are some ethical considerations regarding this study. The patients are already operated, and the planned clinical examination/control poses no risks for the individual patient. The examination is although an extra examination, not a part of any scheduled post-operative check-ups. The examination will take approximately 30 minutes and the patients will not have any obvious advantages by undergoing the examination. During the examination findings might reveal ongoing pathology in some patients. This will be handled accordingly. The examination is also on voluntary basis and all patients included in the original studies were 18 years and older and where able to verify informed consent independently. If a situation will arise where there are doubts regarding a patient's ability to make independent decisions, the patient will not be included in this study.

   If any of the patients eligible for this study still regularly has appointments at the Oral and Maxillofacial unit at Karolinska University Hospital of any kind, they should be ensured that they have the right (as any of the other patients) to not participate in this study, and that this decision will not affect the care given to them in any way.

   Regarding the voluntary radiology examination planned, the patient will be exposed to ionizing radiation with a dose equivalent of 0.2 mSv. Although, there is no radiation dose that is considered as totally harmless, the dose of the planned radiological examination is equivalent with approximately 2,5 month of natural radiation. The average radiation dose in Sweden is approximately 3 mSv/year, and this examination contributes to the patient's total radiation burden. The choice of CBCT and the applied examination protocol is a standard protocol optimized for examination TMJ according to ALARA principle (as low as reasonably achievable). Some patients in the cohort might have an indication for a CBCT because of their symptoms and clinical findings. However, within this project, all the included patients with given consent will be radiologically examined. The examination in itself will possibly not contribute to the well-being of the patient or pose any advantages. On the other hand, unexpected findings might appear that in a wide patient-oriented perspective might be beneficial to detect. The reason that we believe this project justifies performing this radiological examination is the fact that no earlier long-term follow-ups have been presented and that radiological findings, together with the clinical examination, will give a detailed insight into the patient-group´s outcome. This might hypothetically lead to revised follow-up protocols. By identifying potential risk factors, the radiological examinations might be more individualized according to the risk factors of the individual patient. The risk of missing important findings in the CBCT examinations exposed for the study will be low. All the CBCT scans will be examined by a specialist in radiology according to the normal review & referral procedure.
7. RELEVANCE

There are no long-term, prospective, follow-up studies on DD surgery made, as known of. This is why this study will fill a knowledge gap and will lead to new insights in the natural post-operative course of this patient group. This might change how patients are selected for surgery, and perhaps how postoperative follow-ups are scheduled with a more individualized follow up programme.

ELIGIBILITY:
Inclusion Criteria:

* Patients participating in the studies with ethical approval numbers EPN 2014/764-31/2 and 2014/622-31/1.
* Initial diagnosis DDwR or DDwoR.

Exclusion Criteria:

* Patient unable to verify informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort has already been operated (arthroscopy or discectomy) due to temporomandibular joint disc displacement during the years 2014-2017, then participating in a prospective cohort study mainly focusing on surgical outcome predictors (ethical approval: 2014/622-31/1 and 2014/764-31/2). These patients will now be offered a clinical and radiological examination approximately 10 years postoperative.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Treatment success. | From intervention to the 10 year follow up.
  Treatment outcome (successful, good, intermediate, deteriorated). This is ordinal data and a compiled judgement will be made after evaluating four different parameters:
  1. Maximum interincisal opening (MIO) of ≥ 35 mm, or an increase of MIO of ≥ 40 %.
  2. Patient-reported TMJ pain. Visual analogue scale (VAS) ≤ 3, or ≤ 40% reduction.
  3. Patient-reported TMJ disability. VAS ≤ 3, or a 40 % reduction.
  4. Patient-reported TMJ psychosocial impact. VAS ≤ 3, or a 40 % reduction.
     * Successful outcome: criteria 1-4 fulfilled
     * Good: criteria 1 and one or two of criteria 2-4 fulfilled
     * Intermediate: no criterias fulfilled
     * Deteriorated: criterias 1-4 worsened

SECONDARY OUTCOMES:
Joint degeneration | From intervention to the 10 year follow up.
  At the timepoint of long-term examination, a radiological evaluation of the TMJ status will be made with a cone beam computed tomography (CBCT). The patients were evaluated preoperatively with a CBCT scan, which makes it possible to evaluate eventual time dependent deterioration of the joints.

OTHER OUTCOMES:
Maximum interincisal opening | From intervention to the 10 year follow up.
  Measured in millimeters. The distance between teeth 11 and 41 is measured as the patient opens their mouth as wide as possible. If this is not feasible due to malocclusion, tooth loss, etc., an alternative representative pair of front teeth is chosen for measurement. This should be noted in the patient's record to ensure consistent measurements in the future.
Pain in the temporomandibular joint (TMJ) during function | From intervention to the 10 year follow up.
  The patient is asked to estimate how much pain TMJ function (opening, biting, chewing, speaking, etc.) has caused on average over the past 2-week period. This estimation should exclude the worst imaginable pain. Each TMJ is assessed individually, meaning the patient should provide a numerical value between 0 (no pain) and 10 (worst imaginable pain) for each joint.
Pain in the temporomandibular joint at rest | From intervention to the 10 year follow up.
  The patient is asked to estimate pain in each TMJ at rest. The value should reflect an average representative of the past 2-week period.meaning the patient should provide a numerical value between 0 (no pain) and 10 (worst imaginable pain) for each joint.
Functional impairment of the temporomandibular joint | From intervention to the 10 year follow up.
  The patient is asked to estimate the degree of functional impairment caused by current TMJ issues. This variable includes both joint mobility and the ability to consume food. The scale is graded from 0 to 10. A score of 0 indicates no impairment, meaning unrestricted jaw opening and the ability to eat all types of food without difficulty. A score of 10 represents complete functional impairment, such as zero millimeters of opening or being able to consume only liquids due to the inability to chew solid food.
Psychosocial impact | From intervention to the 10 year follow up.
  The patient is asked to estimate the psychosocial impact of their TMJ issues from 0 to 10. A score of 0 indicates no impact, while a score of 10 represents the worst imaginable impact. This may include how much and how often the patient thinks about their TMJ issues, how it affects their mood, and how it impacts their social life, such as withdrawing from social interactions.
Other bodily pain | From intervention to the 10 year follow up.
  The patient is asked to estimate the degree of bodily pain unrelated to TMJ pain between 0 to 10. This can include pain from other joints, gastrointestinal discomfort, etc. A score of 0 indicates no other bodily pain, while a score of 10 indicates the worst imaginable bodily pain.
Palpation tenderness of TMJ | From intervention to the 10 year follow up.
  The TMJ is palpated laterally according to DC/TMD (500 grams pressure). A letter balance is used to calibrate palpation pressure. The pain must be recognizable to the patient.
Palpation tenderness of the masseter and temporalis muscles | From intervention to the 10 year follow up.
  The masseter and temporalis muscles are palpated at three separate sites each, according to DC/TMD (1000 grams pressure). A letter balance is used to calibrate palpation pressure. The pain must be recognizable to the patient.
Maximum protrusion | From intervention to the 10 year follow up.
  Horizontal overbite (HOB) is first measured in millimeters during habitual intercuspal position. The value is positive if tooth 11 is located facially to tooth 41 and negative if the reverse is true. The patient is then instructed to protrude the mandible maximally, and the horizontal distance between the incisal edges of teeth 11 and 41 is measured again. These two measurements are then added together (noting negative HOB in Class III cases).
Maximum laterotrusion | From intervention to the 10 year follow up.
  The patient is instructed to move the mandible to one side. The distance between the midline of the maxilla (between teeth 11 and 21) and the midline of the mandible (between teeth 31 and 41) is measured in millimeters. Any midline deviation during habitual intercuspal position is measured and subtracted from or added to the recorded value. Laterotrusion is measured for both left and right movements.

CONTACTS AND LOCATIONS:
Overall Officials: Mattias Ulmner, DDS, PhD, Principal Investigator — Karolinska Institutet, Department of Dental Medicine
Locations (1):
- Karolinska Institutet, Huddinge, Sweden

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the result published will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and SAP is available through ClinicalTrials.

REFERENCES:
- [Background] Wilkes CH. Internal derangements of the temporomandibular joint. Pathological variations. Arch Otolaryngol Head Neck Surg. 1989 Apr;115(4):469-77. doi: 10.1001/archotol.1989.01860280067019. PMID 2923691
- [Background] Ulmner M, Weiner CK, Lund B. Predictive factors in temporomandibular joint arthroscopy: a prospective cohort short-term outcome study. Int J Oral Maxillofac Surg. 2020 May;49(5):614-620. doi: 10.1016/j.ijom.2019.09.002. Epub 2019 Sep 26. PMID 31564479
- [Background] Ulmner M, Sugars R, Naimi-Akbar A, Tudzarovski N, Kruger-Weiner C, Lund B. Synovial Tissue Proteins and Patient-Specific Variables as Predictive Factors for Temporomandibular Joint Surgery. Diagnostics (Basel). 2020 Dec 30;11(1):46. doi: 10.3390/diagnostics11010046. PMID 33396653
- [Background] Ulmner M, Bjornland T, Rosen A, Berge TI, Olsen-Bergem H, Lund B. Evidence for minimally invasive treatment-A systematic review on surgical management of disc displacement. J Oral Rehabil. 2024 Jun;51(6):1061-1080. doi: 10.1111/joor.13661. Epub 2024 Feb 23. PMID 38400536
- [Background] Sorel B, Piecuch JF. Long-term evaluation following temporomandibular joint arthroscopy with lysis and lavage. Int J Oral Maxillofac Surg. 2000 Aug;29(4):259-63. PMID 11030395
- [Background] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Background] Sale H, Bryndahl F, Isberg A. Temporomandibular joints in asymptomatic and symptomatic nonpatient volunteers: a prospective 15-year follow-up clinical and MR imaging study. Radiology. 2013 Apr;267(1):183-94. doi: 10.1148/radiol.12112243. Epub 2012 Dec 18. PMID 23249569
- [Background] Murakami KI, Tsuboi Y, Bessho K, Yokoe Y, Nishida M, Iizuka T. Outcome of arthroscopic surgery to the temporomandibular joint correlates with stage of internal derangement: five-year follow-up study. Br J Oral Maxillofac Surg. 1998 Feb;36(1):30-4. doi: 10.1016/s0266-4356(98)90744-6. PMID 9578253
- [Background] Murakami K, Segami N, Okamoto M, Yamamura I, Takahashi K, Tsuboi Y. Outcome of arthroscopic surgery for internal derangement of the temporomandibular joint: long-term results covering 10 years. J Craniomaxillofac Surg. 2000 Oct;28(5):264-71. doi: 10.1054/jcms.2000.0162. PMID 11467389
- [Background] Lund B, Ulmner M, Bjornland T, Berge T, Olsen-Bergem H, Rosen A. A disease-focused view on the temporomandibular joint using a Delphi-guided process. J Oral Sci. 2020;62(1):1-8. doi: 10.2334/josnusd.19-0128. PMID 31996510
- [Background] Leibur E, Jagur O, Muursepp P, Veede L, Voog-Oras U. Long-term evaluation of arthroscopic surgery with lysis and lavage of temporomandibular joint disorders. J Craniomaxillofac Surg. 2010 Dec;38(8):615-20. doi: 10.1016/j.jcms.2010.02.003. Epub 2010 Mar 23. PMID 20335040
- [Background] Kircos LT, Ortendahl DA, Mark AS, Arakawa M. Magnetic resonance imaging of the TMJ disc in asymptomatic volunteers. J Oral Maxillofac Surg. 1987 Oct;45(10):852-4. doi: 10.1016/0278-2391(87)90235-7. PMID 3477621
- [Background] Kadesjo N, Benchimol D, Falahat B, Nasstrom K, Shi XQ. Evaluation of the effective dose of cone beam CT and multislice CT for temporomandibular joint examinations at optimized exposure levels. Dentomaxillofac Radiol. 2015;44(8):20150041. doi: 10.1259/dmfr.20150041. Epub 2015 Jun 2. PMID 26119344
- [Background] Ferrillo M, Nucci L, Giudice A, Calafiore D, Marotta N, Minervini G, d'Apuzzo F, Ammendolia A, Perillo L, de Sire A. Efficacy of conservative approaches on pain relief in patients with temporomandibular joint disorders: a systematic review with network meta-analysis. Cranio. 2025 Mar;43(2):258-274. doi: 10.1080/08869634.2022.2126079. Epub 2022 Sep 23. PMID 36148997
- [Background] Eriksson L, Westesson PL. Diskectomy in the treatment of anterior disk displacement of the temporomandibular joint. A clinical and radiologic one-year follow-up study. J Prosthet Dent. 1986 Jan;55(1):106-16. doi: 10.1016/0022-3913(86)90085-5. No abstract available. PMID 3456042
- [Background] Eriksson L, Westesson PL. Long-term evaluation of meniscectomy of the temporomandibular joint. J Oral Maxillofac Surg. 1985 Apr;43(4):263-9. doi: 10.1016/0278-2391(85)90284-8. PMID 3856642
- [Background] Bjornland T, Larheim TA. Discectomy of the temporomandibular joint: 3-year follow-up as a predictor of the 10-year outcome. J Oral Maxillofac Surg. 2003 Jan;61(1):55-60. doi: 10.1053/joms.2003.50010. PMID 12524609
- [Background] Al-Moraissi EA, Wolford LM, Ellis E 3rd, Neff A. The hierarchy of different treatments for arthrogenous temporomandibular disorders: A network meta-analysis of randomized clinical trials. J Craniomaxillofac Surg. 2020 Jan;48(1):9-23. doi: 10.1016/j.jcms.2019.10.004. Epub 2019 Nov 5. PMID 31870713
- [Background] Al-Moraissi EA. Open versus arthroscopic surgery for the management of internal derangement of the temporomandibular joint: a meta-analysis of the literature. Int J Oral Maxillofac Surg. 2015 Jun;44(6):763-70. doi: 10.1016/j.ijom.2015.01.024. Epub 2015 Feb 18. PMID 25701306
- [Background] Al-Moraissi EA. Arthroscopy versus arthrocentesis in the management of internal derangement of the temporomandibular joint: a systematic review and meta-analysis. Int J Oral Maxillofac Surg. 2015 Jan;44(1):104-12. doi: 10.1016/j.ijom.2014.07.008. Epub 2014 Aug 7. PMID 25123511